CLINICAL TRIAL: NCT00126438
Title: An Open-Label, Multicenter, Phase 3 Study Evaluating the Prognostic Usefulness of I-123 mIBG Scintigraphy for Identifying Subjects With Heart Failure Who Will Experience an Adverse Cardiac Event
Brief Title: Meta-Iodobenzylguanidine (123I-mIBG) Scintigraphy Imaging in Patients With Heart Failure and Control Subjects Without Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MBG312
Record Dates: First submitted 2005-08-03; First posted 2005-08-04 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; nuclear cardiology; sympathetic innervation; 123I-mIBG
MeSH Terms: conditions — Heart Failure | interventions — 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 123I-mIBG (meta-iodobenzylguanidine) (Experimental): Single dose
  Interventions: Drug: 123I-mIBG (meta-iodobenzylguanidine)

INTERVENTIONS:
Drug: 123I-mIBG (meta-iodobenzylguanidine) — Single Dose
  Other Names: MIBG; Iobenguane

SUMMARY:
The study is designed to study the utility of 123I-mIBG as a diagnostic imaging agent to predict cardiac outcome in subjects with heart failure and in comparison to subjects without cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must be adults with an established diagnosis of heart failure (New York Heart Association Class II or III) and reduced left ventricular ejection fraction (LVEF) (≤ 35%) or be healthy volunteers without heart disease.

Exclusion Criteria:

* Healthy volunteers were not eligible if they had a history of diabetes mellitus, signs/symptoms of neurological disease (e.g., Parkinson's Disease, multiple system atrophy, Parkinsonian syndromes), or other diseases known to affect the sympathetic nervous system.
* Subjects with New York Heart Association Class I or IV heart failure were not eligible.
* Subjects were excluded if they had previously received 123I-mIBG or 131I-mIBG or participated in a clinical study involving investigational medicinal product or devices within 30 days.
* Subjects that had a pacemaker or had received defibrillation, anti-tachycardia pacing or cardioversion to treat a previous arrhythmic event or had an ICD inserted within 30 days before study entry are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2005-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Strohmeyer, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Hachamovitch R, Nutter B, Menon V, Cerqueira MD. Predicting Risk Versus Predicting Potential Survival Benefit Using 123I-mIBG Imaging in Patients With Systolic Dysfunction Eligible for Implantable Cardiac Defibrillator Implantation: Analysis of Data From the Prospective ADMIRE-HF Study. Circ Cardiovasc Imaging. 2015 Dec;8(12):e003110. doi: 10.1161/CIRCIMAGING.114.003110. PMID 26666380
- [Derived] Gerson MC, Caldwell JH, Ananthasubramaniam K, Clements IP, Henzlova MJ, Amanullah A, Jacobson AF. Influence of diabetes mellitus on prognostic utility of imaging of myocardial sympathetic innervation in heart failure patients. Circ Cardiovasc Imaging. 2011 Mar;4(2):87-93. doi: 10.1161/CIRCIMAGING.110.954784. Epub 2010 Dec 30. PMID 21193691
- [Derived] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 753 participants were screened, of whom 197 were screen failures due to inclusion/exclusion criteria; 24 withdrawn at participant's request; 2 withdrawn at investigator's request and 15 failed to complete all screening procedures.
Pre-assignment Details: A total 515 participants (453 Heart failure [HF] and 62 control) were enrolled in the study and received a single dose of investigational medicinal product (IMP) at 43 investigational centers.
Groups:
- AdreView - Heart Failure Group: AdreView (123I-mIBG [meta-iodobenzylguanidine]): 10 milliCurie (mCi) as a single intravenous dose.
- Adreview - Control Group: AdreView (123I-mIBG): 10 mCi as a single intravenous dose.
Period: Overall Study
Arm/Group | AdreView - Heart Failure Group | Adreview - Control Group
Started | 453 | 62
Completed | 419 | 52
Not Completed | 34 | 10
Not completed — Withdrawal due to adverse event | 1 | 0
Not completed — Lost to Follow-up | 22 | 0
Not completed — Protocol Violation | 8 | 8
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received IMP manufactured by the sponsor.
Groups:
- AdreView - Heart Failure; Adreview - Control Group: AdreView (123I-mIBG): 10 mCi as a single intravenous dose.
- Total: Total of all reporting groups
Arm/Group | AdreView - Heart Failure | Adreview - Control Group | Total
Number analyzed (Participants) | 453 | 62 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.38) | 58.8 (10.84) | 61.2 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 19 | 121
  Male | 351 | 43 | 394

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between the Occurrence of Adverse Cardiac Event and 123I-mIBG Uptake on Planar Scintigraphy Categorized as High or Low Heart to Mediastinum (H/M) Ratio
Description: H/M ratio for 123I-mIBG uptake at 3 hours 50 minutes post administration was calculated by dividing the counts/pixel in the total myocardium region of interest (ROI) by the counts/pixel in the 7x7 pixel mediastinal ROI. Assessments were done by 3 independent readers. H/M ratios were categorized as 'Low' and 'High' based on being <1.6 or ≥1.6 respectively. The efficacy of 123I-mIBG was based on the prognostic value of the imaging data collected relative to time to adverse cardiac events. Data analysis to assess the relative hazard of an adverse cardiac event was performed only on HF participants categorized into 2 groups with H/M <1.6 and H/M ≥1.6 using a Cox proportional hazards model.
Time Frame: Approximately 24 months from the date of administration of 123I-mIBG
Population: Primary efficacy population included 444 participants in HF group who received IMP and had a diagnostic (optimal/sub-optimal) 3 hour 50 minute planar image. Primary efficacy analysis was based on comparing only "Adreview HF" participants with low vs. high H/M and, therefore, did not include "Adreview Control" group.
Measure: Number; unit: number of adverse cardiac events
Groups:
- AdreView-Heart Failure Group With High H/M Ratio: Participants in HF group who had high H/M ratio (more than or equal to 1.6).
- AdreView-Heart Failure Group With Low H/M Ratio: Participants in HF group who had low H/M ratio (less than 1.6).
Arm/Group | AdreView-Heart Failure Group With High H/M Ratio | AdreView-Heart Failure Group With Low H/M Ratio
Number analyzed (Participants) | 86 | 358
number of adverse cardiac events
  Reader A (n=86, 355) | 11 | 111
  Reader B (n=86, 358) | 11 | 113
  Reader C (n=86, 352) | 11 | 112
Statistical Analysis 1: Comparison: AdreView-Heart Failure Group With High H/M Ratio vs AdreView-Heart Failure Group With Low H/M Ratio; Analysis based on Reader A readings. Data analysis to assess the relative hazard of an adverse cardiac event was performed using a Cox proportional hazards model. Hazard (risk) of an event for a participant with low H/M at time "t" was expressed as Hl (t)/ Hh (t) = Ψ, where Hl (t) and Hh (t) denote the hazard of an event at time t for participants with low H/M and high H/M respectively; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Model — At 0.025 level of significance; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.18 to 0.73]
Statistical Analysis 2: Comparison: AdreView-Heart Failure Group With High H/M Ratio vs AdreView-Heart Failure Group With Low H/M Ratio; Analysis based on Reader B readings. Data analysis to assess the relative hazard of an adverse cardiac event was performed using a Cox proportional hazards model. Hazard (risk) of an event for a participant with low H/M at time "t" was expressed as Hl (t)/ Hh (t) = Ψ, where Hl (t) and Hh (t) denote the hazard of an event at time t for participants with low H/M and high H/M respectively; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Model — At 0.025 level of significance; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.18 to 0.72]
Statistical Analysis 3: Comparison: AdreView-Heart Failure Group With High H/M Ratio vs AdreView-Heart Failure Group With Low H/M Ratio; Analysis based on Reader C readings. Data analysis to assess the relative hazard of an adverse cardiac event was performed using a Cox proportional hazards model. Hazard (risk) of an event for a participant with low H/M at time "t" was expressed as Hl (t)/ Hh (t) = Ψ, where Hl (t) and Hh (t) denote the hazard of an event at time t for participants with low H/M and high H/M respectively; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Model — At 0.025 level of significance; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.17 to 0.72]

ADVERSE EVENTS:
Time Frame: Up to 30 hours after administration of the IMP.
Description: Analysis was performed on safety population that included all participants who received a dose of IMP.
Arm/Group | AdreView - Heart Failure | Adreview - Control Group
Serious Adverse Events (participants affected / at risk) | 6/453 | 0/62
Other Adverse Events (participants affected / at risk) | 0/453 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdreView - Heart Failure (N=453) | Adreview - Control Group (N=62)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Pain (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.